CLINICAL TRIAL: NCT00950833
Title: Vaccination Course in Children Primed and Boosted With Pneumococcal Vaccine GSK 1024850A and in Age-matched Unprimed Children
Brief Title: Long-term Follow-up Study of Children Previously Primed With GSK Pneumococcal Vaccine (GSK1024850A) and of Unprimed Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112801
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Infections, Streptococcal
Keywords: Catch-up vaccination; Pneumococcal vaccine; Immune memory; Nasopharyngeal carriage; Immunogenicity; Pneumococcal disease; Safety
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

ARMS (3):
- AP-AP Group (Active Comparator): subjects from the AP-AP group, previously vaccinated with pneumococcal conjugate vaccine GSK1024850A in study NCT00496015, receiving an additional dose of pneumococcal conjugate vaccine GSK1024850A for immune memory assessment
  Interventions: Biological: Pneumococcal vaccine GSK1024850A
- NAP-pre Group (Active Comparator): subjects from the NAP-pre group, previously vaccinated with pneumococcal conjugate vaccine GSK1024850A in study NCT00496015 receiving an additional dose of pneumococcal conjugate vaccine GSK1024850A for immune memory assessment
  Interventions: Biological: Pneumococcal vaccine GSK1024850A
- Unprimed Group (Active Comparator): Age-matched subjects from the unprimed group of the NCT00496015 study, not previously vaccinated with any pneumococcal vaccine, receiving two doses of pneumococcal conjugate vaccine GSK1024850A
  Interventions: Biological: Pneumococcal vaccine GSK1024850A

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — 1 or 2 intramuscular injections

SUMMARY:
The objective of this study is to evaluate the immune memory through the administration of an additional dose of GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A, the antibody persistence and long-term effect on nasopharyngeal carriage of S. pneumoniae and H. influenzae in subjects primed and boosted with GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A in previous primary and booster studies. For subjects that did not receive the investigational vaccine during the primary and booster study, the objective is to evaluate immunogenicity, safety and reactogenicity of a 2-dose catch-up vaccination with GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A.

This protocol posting deals with objectives & outcome measures of the extension phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00370318). The objectives & outcome measures of the booster phase are presented in a separate protocol posting (NCT00496015).

DETAILED DESCRIPTION:
This protocol posting has been updated according to Protocol Amendment 1, July 2009

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/ guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 31 and 34 months of age at the time of the enrolment.
* Subjects who previously participated in study NCT00496015
* For the subjects in the primed AP-AP and NAP-pre groups: subjects who received a booster dose of the pneumococcal conjugate vaccine prior to the study amendment 3.
* For the subjects in the unprimed group: subjects who received a dose of the meningococcal vaccine GSK134612.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding enrolment, or planned use during the entire study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the entire study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of study vaccine and ending 30 days after.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of seizures or progressive neurological disease.
* Acute disease at the time of enrolment, defined as the presence of a mild, moderate or severe illness with or without fever.
* Administration or planned use of immunoglobulins and/ or any blood products during the entire study period.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* Subjects of which both parents have a history of atopia (polinosis, asthma, atopic eczema).
* Administration of any pneumococcal vaccine since the end of study NCT00496015.

Ages: 31 Months to 44 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 466 (Actual)
Dates: Start 2009-08-10 (Actual); Primary Completion 2010-09-16 (Actual); Study Completion 2010-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Czechia (8):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Prymula R, Habib A, Francois N, Borys D, Schuerman L. Immunological memory and nasopharyngeal carriage in 4-year-old children previously primed and boosted with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) with or without concomitant prophylactic paracetamol. Vaccine. 2013 Apr 12;31(16):2080-8. doi: 10.1016/j.vaccine.2013.01.044. Epub 2013 Feb 5. PMID 23391599
- [Background] Prymula R et al. Immune memory 2-3 years after vaccination with pneumococcal non-typeable Heamophilus influenzae protein-D conjugate vaccine (PHiD-CV), with or without prophylactic paracetamol. Abstract presented at the 30th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID), Thessaloniki, Greece, 8-12 May 2012.
- [Background] Prymula R et al. Long-term effect of 10-valent pneumococcal non-typeable Haemophilus Influenzae protein D conjugate vaccine (PHiD-CV) on nasopharyngeal bacterial carriage in Czech children. Abstract presented at the 8th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Iguaçu Falls, Brazil, 11-15 March, 2012.
- [Background] Silfverdal SA et al. Immunogenicity and reactogenicity of 2-dose catch-up vaccination with 10-valent pneumococcal non-typeable Haemophilus Influenzae protein D conjugate vaccine (PHiD-CV) during the fourth year of life. Abstract presented at the 8th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD), Iguaçu Falls, Brazil, 11-15 March, 2012.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 466 subjects enrolled in the study, 5 subjects were not included in the Total effective cohort as they did not meet eligibility criteria. Out of the 461 subjects enrolled in the Total effective cohort, 18 subjects were not included in the Total vaccinated cohort as these subjects withdrew before the first vaccination visit (Visit 2).
Groups:
- Synflorix I Group: Healthy male or female subjects between and including 31 and 44 months of age at the time of enrolment, who were previously given 3 primary vaccination doses of Synflorix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107017 (NCT00370318) and one booster dose of Synflorix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107137 (NCT00496015), additionally received in the current study one dose of Synflorix™ vaccine at Month 9 (40-48 months of age), administered intramuscularly in the deltoid muscle. At the time of both primary and booster vaccinations, subjects received prophylactic antipyretic (AP) treatment with paracetamol.
- Synflorix II Group: Healthy male or female subjects between and including 31 and 44 months of age at the time of enrolment, who were previously given 3 primary vaccination doses of Synflorix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107017 (NCT00370318) and one booster dose of Synflorix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107137 (NCT00496015), additionally received in the current study one dose of Synflorix™ vaccine at Month 9 (40-48 months of age), administered intramuscularly in the deltoid muscle. At the time of both primary and booster vaccinations, subjects did not receive any prophylactic antipyretic (AP) treatment.
- Synflorix III Group: Healthy male or female subjects between and including 31 and 44 months of age at the time of enrolment, who were not previously primed with Synflorix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107137 (NCT00496015), but vaccinated with Nimenrix™ vaccine co-administered with Infanrix™ Hexa vaccine in study 107137 (NCT00496015), additionally received in the current study 2 doses of Synflorix™ vaccine at Month 9 (40-48 months of age) and at Month 11 (42-50 months of age), administered intramuscularly in the deltoid muscle.
Period: Overall Study
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group
Started | 112 | 108 | 223
Completed | 112 | 108 | 223
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group | Total
Number analyzed (Participants) | 112 | 108 | 223 | 443
Age, Continuous [Mean (Standard Deviation); unit: Months] | 39.2 (1.53) | 39.1 (1.54) | 37.7 (3.36) | 38.4 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 48 | 99 | 207
  Male | 52 | 60 | 124 | 236
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European heritage | 111 | 108 | 214 | 433
  White - Arabic / North African heritage | 0 | 0 | 9 | 9
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: Antibody concentrations against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) have been assessed by 22F-inhibition enzyme linked immunosorbent assay (ELISA), presented as geometric mean concentrations (GMCs) and expressed in micrograms per milliliter (μg/mL). The seropositivity cut-off value of the assay was an antibody concentration greater than or equal to (≥) 0.05 μg/mL.
Time Frame: At 7-10 days after the first vaccine dose
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one pneumococcal vaccine serotype were available after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- Pooled Synflorix I+II Group: For the purpose of the analysis, subjects from Synflorix I Group and Synflorix II Group have been pooled into a sub-group.
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 204 | 215
μg/mL
  Anti-1 | 1.24 [1.07 to 1.42] | 7.63 [6.57 to 8.86]
  Anti-4 | 4.52 [3.96 to 5.17] | 12.95 [11.37 to 14.75]
  Anti-5: number analyzed (Participants) | 202 | 215
  Anti-5 | 0.72 [0.63 to 0.84] | 9.76 [8.44 to 11.29]
  Anti-6B: number analyzed (Participants) | 203 | 215
  Anti-6B | 0.27 [0.22 to 0.33] | 7.67 [6.7 to 8.78]
  Anti-7F | 1.37 [1.19 to 1.58] | 6.51 [5.69 to 7.46]
  Anti-9V: number analyzed (Participants) | 202 | 213
  Anti-9V | 0.69 [0.58 to 0.83] | 9.75 [8.46 to 11.24]
  Anti-14: number analyzed (Participants) | 204 | 214
  Anti-14 | 1.01 [0.8 to 1.27] | 23.07 [20.03 to 26.57]
  Anti-18C: number analyzed (Participants) | 204 | 214
  Anti-18C | 3.25 [2.71 to 3.9] | 32.54 [28.15 to 37.61]
  Anti-19F: number analyzed (Participants) | 204 | 214
  Anti-19F | 4.31 [3.59 to 5.17] | 39.84 [34.12 to 46.51]
  Anti-23F | 0.25 [0.2 to 0.32] | 9.24 [7.86 to 10.86]
Statistical Analysis 1: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory induced for anti-pneumococcal serotype 1 following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 1; ANOVA; GMC ratio for anti-1 = 6.17, 95% CI 2-sided [5.03 to 7.58]
Statistical Analysis 2: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 4 induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled SynflorixI+II Group over Synflorix Group) was higher than 1 for pneumococcal serotype 4; ANOVA; GMC ratio for anti-4 = 2.86, 95% CI 2-sided [2.38 to 3.45]
Statistical Analysis 3: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 5 induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 5; ANOVA; GMC ratio for anti-5 = 13.47, 95% CI 2-sided [10.96 to 16.55]
Statistical Analysis 4: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 6B induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 6B; ANOVA; GMC ratio for anti-6B = 28.81, 95% CI 2-sided [22.54 to 36.81]
Statistical Analysis 5: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 7F induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 7F; ANOVA; GMC ratio for anti-7F = 4.75, 95% CI 2-sided [3.9 to 5.78]
Statistical Analysis 6: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 9V induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 9V; ANOVA; GMC ratio for anti-9V = 14.1, 95% CI 2-sided [11.21 to 17.75]
Statistical Analysis 7: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 14 induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 14; ANOVA; GMC ratio for anti-14 = 22.92, 95% CI 2-sided [17.51 to 30]
Statistical Analysis 8: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 18C induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 18C; ANOVA; GMC ratio for anti-18C = 10.01, 95% CI 2-sided [7.95 to 12.61]
Statistical Analysis 9: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 19F induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 19F; ANOVA; GMC ratio for anti-19F = 9.25, 95% CI 2-sided [7.29 to 11.74]
Statistical Analysis 10: Comparison: Synflorix III Group vs Pooled Synflorix I+II Group; To demonstrate the immunological memory for anti-pneumococcal serotype 23F induced following primary vaccination in study 107017 (NCT00370318) and booster vaccination in study 107137 (NCT00496015) with the Synflorix™ vaccine, through evaluation of early antibody responses after an additional dose of Synflorix™ vaccine at 40-48 months of age, compared to the Synflorix III Group; Test type: Non-Inferiority — The immune memory would be demonstrated if the lower limit (LL) of the 95% confidence interval (CI) around the geometric mean concentration (GMC) ratios (Pooled Synflorix I+II Group over Synflorix III Group) was higher than 1 for pneumococcal serotype 23F; ANOVA; GMC ratio for anti-23F = 36.52, 95% CI 2-sided [27.59 to 48.34]

2. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: Antibody concentrations against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) have been assessed by 22F-inhibition ELISA, presented as GMCs and expressed in μg/mL. The seropositivity cut-off value of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: Prior to the first study vaccine dose (At Day 0)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against at least one pneumococcal vaccine serotype were available after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 209 | 215
μg/mL
  Anti-1: number analyzed (Participants) | 208 | 215
  Anti-1 | 0.09 [0.08 to 0.11] | 0.27 [0.23 to 0.33]
  Anti-4: number analyzed (Participants) | 206 | 213
  Anti-4 | 0.05 [0.04 to 0.06] | 0.2 [0.17 to 0.23]
  Anti-5: number analyzed (Participants) | 208 | 212
  Anti-5 | 0.1 [0.09 to 0.11] | 0.41 [0.36 to 0.47]
  Anti-6B: number analyzed (Participants) | 202 | 212
  Anti-6B | 0.1 [0.08 to 0.12] | 0.8 [0.61 to 1.05]
  Anti-7F | 0.06 [0.05 to 0.07] | 0.48 [0.41 to 0.56]
  Anti-9V: number analyzed (Participants) | 203 | 211
  Anti-9V | 0.07 [0.06 to 0.09] | 0.5 [0.41 to 0.61]
  Anti-14: number analyzed (Participants) | 203 | 213
  Anti-14 | 0.28 [0.22 to 0.36] | 1.21 [0.97 to 1.5]
  Anti-18C: number analyzed (Participants) | 205 | 215
  Anti-18C | 0.09 [0.07 to 0.11] | 0.65 [0.54 to 0.79]
  Anti-19F: number analyzed (Participants) | 208 | 215
  Anti-19F | 0.44 [0.32 to 0.59] | 2.35 [1.75 to 3.15]
  Anti-23F: number analyzed (Participants) | 207 | 215
  Anti-23F | 0.08 [0.07 to 0.1] | 0.96 [0.72 to 1.29]

3. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Vaccine Pneumococcal Serotypes
Description: Seropositivity status was defined as the opsonophagocytic activity (OPA) against pneumococcal serotypes ≥ the value of 8, presented as geometric mean titers (GMTs). The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F).
Time Frame: Prior to (Day 0) and 7-10 days after the first vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 191 | 199
Titers
  Opsono-1, D0 | 5.4 [4.7 to 6.2] | 10.2 [8 to 12.9]
  Opsono-1, D7-10: number analyzed (Participants) | 182 | 194
  Opsono-1, D7-10 | 632 [524.4 to 761.7] | 3106.5 [2670 to 3614.5]
  Opsono-4, D0: number analyzed (Participants) | 174 | 189
  Opsono-4, D0 | 9.1 [6.8 to 12.1] | 18.1 [13.1 to 24.9]
  Opsono-4, D7-10: number analyzed (Participants) | 187 | 195
  Opsono-4, D7-10 | 13109.9 [11080.6 to 15510.7] | 27273.3 [22682.9 to 32792.6]
  Opsono-5, D0: number analyzed (Participants) | 185 | 199
  Opsono-5, D0 | 4 [4 to 4.1] | 8.9 [7.6 to 10.5]
  Opsono-5, D7-10: number analyzed (Participants) | 182 | 194
  Opsono-5, D7-10 | 145.8 [111.7 to 190.3] | 1020 [874 to 1190.2]
  Opsono-6B, D0: number analyzed (Participants) | 173 | 183
  Opsono-6B, D0 | 46.7 [29.8 to 73.3] | 163.5 [108.5 to 246.4]
  Opsono-6B, D7-10: number analyzed (Participants) | 184 | 192
  Opsono-6B, D7-10 | 1472.2 [1053.2 to 2057.8] | 5789.5 [4637.3 to 7227.9]
  Opsono-7F, D0: number analyzed (Participants) | 167 | 187
  Opsono-7F, D0 | 973.4 [798.5 to 1186.6] | 1112.3 [951.4 to 1300.4]
  Opsono-7F, D7-10: number analyzed (Participants) | 186 | 191
  Opsono-7F, D7-10 | 13647.4 [11801.9 to 15781.3] | 19988.9 [16834.5 to 23734.2]
  Opsono-9V, D0: number analyzed (Participants) | 156 | 171
  Opsono-9V, D0 | 268.2 [192.2 to 374.3] | 481.8 [394.6 to 588.1]
  Opsono-9V, D7-10: number analyzed (Participants) | 186 | 194
  Opsono-9V, D7-10 | 14668.8 [12476.1 to 17247] | 17952.5 [14699.2 to 21925.7]
  Opsono-14, D0: number analyzed (Participants) | 166 | 184
  Opsono-14, D0 | 145.3 [97.5 to 216.6] | 267.6 [196.9 to 363.8]
  Opsono-14, D7-10: number analyzed (Participants) | 187 | 195
  Opsono-14, D7-10 | 4454.3 [3921.1 to 5059.9] | 16256.8 [13573 to 19471.4]
  Opsono-18C, D0: number analyzed (Participants) | 169 | 186
  Opsono-18C, D0 | 5.7 [4.7 to 7] | 14.2 [10.6 to 19.2]
  Opsono-18C, D7-10: number analyzed (Participants) | 180 | 188
  Opsono-18C, D7-10 | 9092.2 [7381.2 to 11199.9] | 7413.8 [6072.3 to 9051.6]
  Opsono-19F, D0: number analyzed (Participants) | 186 | 192
  Opsono-19F, D0 | 12.9 [9.6 to 17.2] | 79.5 [55.4 to 113.9]
  Opsono-19F, D7-10: number analyzed (Participants) | 190 | 192
  Opsono-19F, D7-10 | 902.5 [659.2 to 1235.6] | 6271.1 [4814.8 to 8168]
  Opsono-23F, D0: number analyzed (Participants) | 166 | 189
  Opsono-23F, D0 | 220.6 [132 to 368.7] | 462.7 [292.9 to 730.9]
  Opsono-23F, D7-10: number analyzed (Participants) | 189 | 197
  Opsono-23F, D7-10 | 5776.5 [4686.8 to 7119.5] | 15613.5 [12386.9 to 19680.6]

4. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: The vaccine pneumococcal cross-reactive serotypes 6A and 19A have been assessed by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs) and expressed in μg/mL. The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: Prior to (Day 0) and 7-10 days after the first vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 207 | 215
μg/mL
  Anti-6A, D0: number analyzed (Participants) | 207 | 214
  Anti-6A, D0 | 0.11 [0.09 to 0.13] | 0.39 [0.3 to 0.5]
  Anti-6A, D7-10: number analyzed (Participants) | 203 | 215
  Anti-6A, D7-10 | 0.2 [0.17 to 0.25] | 2.4 [2.01 to 2.85]
  Anti-19A, D0 | 0.22 [0.18 to 0.28] | 0.52 [0.41 to 0.67]
  Anti-19A, D7-10: number analyzed (Participants) | 203 | 214
  Anti-19A, D7-10 | 0.65 [0.52 to 0.82] | 6.75 [5.41 to 8.41]

5. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: Seropositivity status was defined as the opsonophagocytic activity against pneumococcal cross-reactive serotypes 6A and 19A (Opsono-16A and opsono-19A) ≥ the value of 8, presented as geometric mean titers (GMTs).
Time Frame: Prior to (Day 0) and 7-10 days after the first vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 183 | 191
Titers
  Opsono-6A, D0: number analyzed (Participants) | 167 | 178
  Opsono-6A, D0 | 49 [32.4 to 74] | 95.2 [65.3 to 138.7]
  Opsono-6A, D7-10: number analyzed (Participants) | 180 | 191
  Opsono-6A, D7-10 | 863.3 [619.3 to 1203.4] | 2408.4 [1815.7 to 3194.5]
  Opsono-19A, D0: number analyzed (Participants) | 183 | 190
  Opsono-19A, D0 | 10.3 [7.9 to 13.4] | 15.9 [11.7 to 21.6]
  Opsono-19A, D7-10: number analyzed (Participants) | 175 | 191
  Opsono-19A, D7-10 | 880.5 [622.7 to 1245] | 2104.9 [1560.9 to 2838.7]

6. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: Anti-protein D (anti-PD) concentrations were presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL). The seropositivity cut-off value of the assay was an antibody concentration ≥ 100 EL.U/mL.
Time Frame: Prior to (Day 0) and 7-10 days after the first vaccine dose
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures and assay results for antibodies against protein D were available after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 204 | 215
EL.U/mL
  Anti-PD, D0: number analyzed (Participants) | 198 | 210
  Anti-PD, D0 | 105.6 [93.8 to 119] | 464.2 [401.6 to 536.5]
  Anti-PD, D7-10 | 374.3 [315.1 to 444.6] | 2673.7 [2359.1 to 3030.2]

7. Secondary Outcome: Memory B-cell Detection for Vaccine Polysaccharides (PS)
Description: B-cell detection for the pneumococcal serotype specific polysaccharides (1, 5, 6B, 18C, 19F, 23F and C) was tabulated for a subset of subjects from each group. The results are expressed as the frequencies of antigen-specific memory B-cells within the total memory B-cell population.
Time Frame: Prior to (Day 0) and 7-10 days after the first vaccine dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Memory B-cells
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group
Number analyzed (Participants) | 70 | 71 | 133
Memory B-cells
  1 PS, D0: number analyzed (Participants) | 23 | 22 | 47
  1 PS, D0 | 288.6 (352.5) | 269.5 (432.2) | 254.8 (368.4)
  1 PS, D7-10: number analyzed (Participants) | 23 | 23 | 43
  1 PS, D7-10 | 1488.8 (1584.2) | 1017.4 (1309.9) | 755.9 (1017.4)
  5 PS, D0: number analyzed (Participants) | 26 | 27 | 42
  5 PS, D0 | 139.4 (214.7) | 141.9 (232.4) | 81.5 (109.2)
  5 PS, D7-10: number analyzed (Participants) | 28 | 23 | 37
  5 PS, D7-10 | 233.5 (235.7) | 406.6 (447.8) | 152.6 (231)
  6B PS, D0: number analyzed (Participants) | 20 | 22 | 44
  6B PS, D0 | 372 (545.5) | 327.2 (554.4) | 639.9 (846.5)
  6B PS, D7-10: number analyzed (Participants) | 16 | 24 | 42
  6B PS, D7-10 | 629.1 (773.2) | 1265.8 (1738.6) | 526 (648.6)
  18C PS, D0: number analyzed (Participants) | 26 | 26 | 42
  18C PS, D0 | 537.7 (641.8) | 530.9 (693.8) | 135.2 (200.6)
  18C PS, D7-10: number analyzed (Participants) | 28 | 23 | 36
  18C PS, D7-10 | 3839 (5960.5) | 8308.4 (7166.9) | 2053.8 (2122.2)
  19F PS, D0: number analyzed (Participants) | 20 | 22 | 44
  19F PS, D0 | 169.7 (415.3) | 149.1 (194.4) | 164.5 (343.4)
  19F PS, D7-10: number analyzed (Participants) | 16 | 23 | 42
  19F PS, D7-10 | 1056.7 (1334) | 1092.4 (1724.3) | 708.2 (1609.4)
  23F PS, D0: number analyzed (Participants) | 23 | 22 | 45
  23F PS, D0 | 112.6 (176.1) | 285 (484.3) | 185.6 (270.1)
  23F PS, D7-10: number analyzed (Participants) | 23 | 23 | 43
  23F PS, D7-10 | 579.8 (632.5) | 1123.7 (2095.4) | 327.9 (470.5)
  C-PS, D0 | 475.9 (682.3) | 462.5 (704.5) | 469.9 (639.2)
  C-PS, D7-10: number analyzed (Participants) | 67 | 70 | 123
  C-PS, D7-10 | 679.2 (885.8) | 915.5 (1191.3) | 762.6 (1039.4)

8. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Serotypes
Description: The vaccine pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F-inhibition ELISA, presented as geometric mean concentrations (GMCs), expressed in μg/mL. The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 μg/mL.
Time Frame: At Month 12, one month after the second vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 209
μg/mL
  Anti-1 | 2.33 [2.13 to 2.54]
  Anti-4 | 6.26 [5.73 to 6.84]
  Anti-5 | 2.69 [2.44 to 2.96]
  Anti-6B | 0.84 [0.73 to 0.97]
  Anti-7F: number analyzed (Participants) | 208
  Anti-7F | 3.63 [3.33 to 3.95]
  Anti-9V | 1.73 [1.56 to 1.93]
  Anti-14 | 5.21 [4.6 to 5.89]
  Anti-18C | 13.59 [11.91 to 15.51]
  Anti-19F | 11.83 [10.35 to 13.52]
  Anti-23F | 0.99 [0.86 to 1.15]

9. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Vaccine Pneumococcal Serotypes
Description: as for outcome 3
Time Frame: At Month 12, one month after the second vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 201
Titers
  Opsono-1 | 125.6 [105 to 150.1]
  Opsono-4: number analyzed (Participants) | 200
  Opsono-4 | 2451.2 [2203.6 to 2726.8]
  Opsono-5: number analyzed (Participants) | 198
  Opsono-5 | 57.2 [47.3 to 69.1]
  Opsono-6B: number analyzed (Participants) | 196
  Opsono-6B | 1345 [1066.8 to 1695.7]
  Opsono-7F: number analyzed (Participants) | 198
  Opsono-7F | 6527.2 [5836.5 to 7299.6]
  Opsono-9V: number analyzed (Participants) | 197
  Opsono-9V | 6091.6 [5328.7 to 6963.8]
  Opsono-14: number analyzed (Participants) | 197
  Opsono-14 | 4544.9 [4030.2 to 5125.4]
  Opsono-18C: number analyzed (Participants) | 196
  Opsono-18C | 3827.5 [3367.5 to 4350.4]
  Opsono-19F | 1251 [1045.6 to 1496.8]
  Opsono-23F: number analyzed (Participants) | 198
  Opsono-23F | 4629.1 [3890.6 to 5507.8]

10. Secondary Outcome: Antibody Concentrations Against Vaccine Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: as for outcome 4
Time Frame: At Month 12, one month after the second vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 209
μg/mL
  Anti-6A | 0.51 [0.43 to 0.6]
  Anti-19A | 1.99 [1.68 to 2.36]

11. Secondary Outcome: Opsonophagocytic Activity (OPA) Titers Against Pneumococcal Cross-reactive Serotypes 6A and 19A
Description: as for outcome 5
Time Frame: At Month 12, one month after the second vaccine dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 196
Titers
  Opsono-6A: number analyzed (Participants) | 193
  Opsono-6A | 918.6 [742.7 to 1136.1]
  Opsono-19A | 597.6 [467.2 to 764.4]

12. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD)
Description: as for outcome 6
Time Frame: At Month 12, one month after the second vaccine dose
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 209
EL.U/mL | 785.9 [695.7 to 887.7]

13. Secondary Outcome: Rabbit Complement-mediated Serum Bactericidal Activity Titers Against Neisseria Meningitidis Serogroups (rSBA-Men)
Description: The Neisseria meningitidis serogroups assessed using rabbit complement were: A, C, W-135 and Y (rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY), presented as geometric mean titers (GMTs). The seropositivity cut-off of the assay was an antibody titer ≥ 8.
Time Frame: At 25-36 months post-vaccination in previous 107137 (NCT00496015) study
Population: The analysis was performed on the ATP cohort for antibody persistence, which included all subjects with the vaccine administration documented, for whom assay results were available for antibodies against each considered antigen for the blood sample taken before the administration of Synflorix™ vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 83
Titers
  rSBA-MenA: number analyzed (Participants) | 66
  rSBA-MenA | 325.5 [243.9 to 434.5]
  rSBA-MenC: number analyzed (Participants) | 80
  rSBA-MenC | 63.6 [41.2 to 98]
  rSBA-MenY | 372.2 [270 to 513]
  rSBA-MenW-135 | 247.6 [190.7 to 321.5]

14. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site. This outcome measure refers only to the primed groups.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 112 | 108
Participants
  Any Pain | 75 | 67
  Grade 3 Pain | 7 | 5
  Any Redness | 58 | 60
  Grade 3 Redness | 13 | 12
  Any Swelling | 43 | 41
  Grade 3 Swelling | 11 | 11

15. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site. This outcome measure refers only to the unprimed group.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 223
Participants
  Any pain, D1 | 150
  Grade 3 pain, D1 | 13
  Any redness, D1 | 102
  Grade 3 redness, D1 | 23
  Any swelling, D1 | 78
  Grade 3 swelling, D1 | 14
  Any pain, D2: number analyzed (Participants) | 222
  Any pain, D2 | 121
  Grade 3 pain, D2: number analyzed (Participants) | 222
  Grade 3 pain, D2 | 12
  Any redness, D2: number analyzed (Participants) | 222
  Any redness, D2 | 93
  Grade 3 redness, D2: number analyzed (Participants) | 222
  Grade 3 redness, D2 | 12
  Any swelling, D2: number analyzed (Participants) | 222
  Any swelling, D2 | 65
  Grade 3 swelling, D2: number analyzed (Participants) | 222
  Grade 3 swelling, D2 | 3
  Any pain, Across doses | 167
  Grade 3 pain, Across doses | 23
  Any redness, Across doses | 127
  Grade 3 redness, Across doses | 29
  Any swelling, Across doses | 101
  Grade 3 swelling, Across doses | 16

16. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as causally related to study vaccination. This outcome measure refers only to the primed groups.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group
Number analyzed (Participants) | 112 | 108
Participants
  Any drowsiness | 41 | 34
  Grade 3 drowsiness | 0 | 0
  Related drowsiness | 26 | 26
  Any Irritability | 33 | 26
  Grade 3 Irritability | 1 | 0
  Related Irritability | 21 | 16
  Any loss of appetite | 23 | 15
  Grade 3 loss of appetite | 1 | 1
  Related loss of appetite | 13 | 10
  Any fever (Axillary) | 12 | 8
  Grade 3 fever (Axillary) | 0 | 1
  Related fever | 10 | 5

17. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as causally related to study vaccination. This outcome measure refers only to the unprimed group.
Time Frame: During the 4-day (Days 0-3) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group
Number analyzed (Participants) | 223
Participants
  Any drowsiness, D1 | 79
  Grade 3 drowsiness, D1 | 1
  Related drowsiness, D1 | 56
  Any Irritability, D1 | 69
  Grade 3 Irritability, D1 | 2
  Related irritability, D1 | 49
  Any loss of appetite, D1 | 47
  Grade 3 loss of appetite, D1 | 5
  Related loss of appetite, D1 | 32
  Any fever (Axillary), D1 | 23
  Grade 3 fever (Axillary), D1 | 1
  Related fever, D1 | 15
  Any drowsiness, D2: number analyzed (Participants) | 222
  Any drowsiness, D2 | 60
  Grade 3 drowsiness, D2: number analyzed (Participants) | 222
  Grade 3 drowsiness, D2 | 1
  Related drowsiness, D2: number analyzed (Participants) | 222
  Related drowsiness, D2 | 43
  Any Irritability, D2: number analyzed (Participants) | 222
  Any Irritability, D2 | 59
  Grade 3 Irritability, D2: number analyzed (Participants) | 222
  Grade 3 Irritability, D2 | 1
  Related irritability, D2: number analyzed (Participants) | 222
  Related irritability, D2 | 44
  Any loss of appetite, D2: number analyzed (Participants) | 222
  Any loss of appetite, D2 | 26
  Grade 3 loss of appetite, D2: number analyzed (Participants) | 222
  Grade 3 loss of appetite, D2 | 1
  Related loss of appetite, D2: number analyzed (Participants) | 222
  Related loss of appetite, D2 | 16
  Any fever (Axillary), D2: number analyzed (Participants) | 222
  Any fever (Axillary), D2 | 9
  Grade 3 fever (Axillary), D2: number analyzed (Participants) | 222
  Grade 3 fever (Axillary), D2 | 1
  Related fever, D2: number analyzed (Participants) | 222
  Related fever, D2 | 5
  Any drowsiness, Across doses | 102
  Grade 3 drowsiness, Across doses | 2
  Related drowsiness, Across doses | 73
  Any Irritability, Across doses | 98
  Grade 3 Irritability, Across doses | 3
  Related irritability, Across doses | 74
  Any loss of appetite, Across doses | 61
  Grade 3 loss of appetite, Across doses | 6
  Related loss of appetite, Across doses | 42
  Any fever (Axillary), Across doses | 30
  Grade 3 fever (Axillary), Across doses | 2
  Related fever, Across doses | 19

18. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Days 0-30) after each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group
Number analyzed (Participants) | 112 | 108 | 223
Participants | 24 | 29 | 73

19. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Month 10 or Month 12)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group
Number analyzed (Participants) | 112 | 108 | 223
Participants | 0 | 0 | 0

20. Secondary Outcome: Number of Nasopharyngeal Swabs With Streptococcus Pneumoniae (Vaccine Serotypes)
Description: Positive cultures of S. pneumoniae Synflorix™ vaccine serotypes identified in the nasopharynx were recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: The analysis was performed on the ATP cohort for carriage, which included all evaluable subjects for whom carriage outcome measures were available after the swab time point.
Measure: Number; unit: Swabs associated to specified bacteria
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Swabs associated to specified bacteria
  31-44 months | 40 | 21
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 46 | 20

21. Secondary Outcome: Number of Nasopharyngeal Swabs With S.Pneumoniae (Cross-reactive Serotypes)
Description: Positive cultures of S. pneumoniae cross- reactive serotypes identified in the nasopharynx were recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Number; unit: Swabs associated to specified bacteria
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Swabs associated to specified bacteria
  31-44 months | 9 | 13
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 19 | 18

22. Secondary Outcome: Number of Nasopharyngeal Swabs With S.Pneumoniae (Non-vaccine and Non-cross-reactive Serotypes)
Description: Positive cultures of S. pneumoniae non- Synflorix™ vaccine, non-cross-reactive serotypes identified in the nasopharynx were recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Number; unit: Swabs associated to specified bacteria
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Swabs associated to specified bacteria
  31-44 months | 25 | 34
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 27 | 35

23. Secondary Outcome: Number of Nasopharyngeal Swabs With Haemophilus Influenzae
Description: Positive cultures of H. influenzae identified in the nasopharynx were recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Number; unit: Swabs associated to specified bacteria
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Swabs associated to specified bacteria
  31-44 months | 43 | 54
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 89 | 74

24. Secondary Outcome: Number of Subjects With New Acquisition of S. Pneumoniae (Vaccine Serotypes) in Nasopharyngeal Swabs
Description: The number of subjects with new acquisition of S. pneumoniae (Synflorix™ vaccine serotypes) detected in nasopharyngeal swabs was recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Participants
  31-44 months | 39 | 20
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 41 | 18

25. Secondary Outcome: Number of Subjects With New Acquisition of S. Pneumoniae (Cross-reactive Serotypes) in Nasopharyngeal Swabs
Description: The number of subjects with new acquisition of S. pneumoniae (cross-reactive serotypes) detected in nasopharyngeal swabs was recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Participants
  31-44 months | 9 | 13
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 18 | 18

26. Secondary Outcome: Number of Subjects With New Acquisition of S. Pneumoniae (Non-vaccine and Non-cross-reactive Serotypes) in Nasopharyngeal Swabs
Description: The number of subjects with new acquisition of S. pneumoniae (non-vaccine and non-cross-reactive serotypes) detected in nasopharyngeal swabs was recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Participants
  31-44 months | 24 | 32
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 25 | 33

27. Secondary Outcome: Number of Subjects With New Acquisition of H. Influenzae in Nasopharyngeal Swabs
Description: The number of subjects with new acquisition of H. influenzae detected in nasopharyngeal swabs was recorded.
Time Frame: At 31-44 months of age and prior to the first vaccine dose, at 40-48 months of age
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix III Group | Pooled Synflorix I+II Group
Number analyzed (Participants) | 210 | 216
Participants
  31-44 months | 35 | 49
  40-48 months: number analyzed (Participants) | 208 | 212
  40-48 months | 70 | 50

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) follow-up periods after vaccination. Unsolicited AEs: within the 31-day (Days 0-30) follow-up periods after vaccination. SAEs: during the entire study period (from Day 0 up to Month 10/12).
Arm/Group | Synflorix I Group | Synflorix II Group | Synflorix III Group
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/108 | 0/223
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/108 | 0/223
Other Adverse Events (participants affected / at risk) | 96/112 | 86/108 | 190/223
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix I Group (N=112) | Synflorix II Group (N=108) | Synflorix III Group (N=223)
Pain (General disorders) | 75 | 67 | 167
Redness (General disorders) | 58 | 60 | 127
Swelling (General disorders) | 43 | 41 | 101
Drowsiness (General disorders) | 41 | 34 | 102
Irritability (General disorders) | 33 | 26 | 98
Loss of appetite (General disorders) | 23 | 15 | 61
Fever/(Axillary) (General disorders) | 12 | 8 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.